CLINICAL TRIAL: NCT01258712
Title: Randomized, Placebo-controlled Study of Tocilizumab in Combination With Methotrexate for Treatment of Moderate to Severe Rheumatoid Arthritis Patients
Brief Title: Study of Tocilizumab in Combination With Methotrexate for Treatment of Moderate to Severe Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharma Taiwan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRA230TW
Record Dates: First submitted 2010-12-08; First posted 2010-12-13 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Tocilizumab + methotrexate(MTX)
- 2 (Placebo Comparator)
  Interventions: Drug: Tocilizumab placebo + methotrexate(MTX)

INTERVENTIONS:
Drug: Tocilizumab + methotrexate(MTX) — Tocilizumab:8 mg/kg every4weeks,IV infusion methotrexate:10-20 mg/week
  Arms: 1
Drug: Tocilizumab placebo + methotrexate(MTX) — Tocilizumab placebo:8 mg/kg every 4 weeks,IV infusion methotrexate:10-20 mg/week
  Arms: 2

SUMMARY:
This is a Phase III study to evaluate efficacy and safety of Tocilizumab in patients with Rheumatoid Arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with history of moderate-to- severe rheumatoid arthritis for more than 6 months according to the American College of Rheumatology (ACR) 1987 revised criteria for the classification of RA.
* Patients who failed to achieve clinical response to treatment of at least 2 DMARDs(disease modifying anti-rheumatic drug) (including MTX) for at least 12 weeks within 12 months prior to screening, of which MTX must have been at a stable dose of 10-20 mg/wk for at least 12 weeks prior to screening. All other DMARDs should be given at standard therapeutic dose.
* Patients who satisfy swollen joint count (SJC) ≥ 6 (66 joint count) and tender joint count (TJC) ≥ 8 (68 joint count) at screening and baseline.
* C-reactive protein (CRP) level ≥ 1 mg/dl or an erythrocyte sedimentation rate (ESR) ≥ 28 mm/hour at screening and at baseline.

Exclusion Criteria:

* Patients who have received a major surgery including joint surgery 8 weeks prior to the screening or are scheduled to be operated within 6 months after the enrolment.
* Patients with rheumatoid autoimmune disease other than RA, including but not limited to SLE(system lupus erythematosus), or significant systemic involvement secondary to RA.
* Patients who belong to the Class IV of the ACR classification criteria for functional status of RA. (ACR Amended Criteria for the Classification of Functional Capacity in Rheumatoid Arthritis; Class IV: Largely or wholly incapacitated with patient bedridden or confined to wheel chair, permitting little or no self-care).
* Patients with a history of hypersensitivity to human, humanized or murine monoclonal antibodies or patients with contraindication for them.
* Patients who currently have or have a history of recurrence of bacterial, viral,fungal, or mycobacterial infections or other infectious diseases; tuberculosis(TB),atypical mycobacterial disease, clinically significant granulomatous disease on chest radiograph, hepatitis B, hepatitis C, or herpes zoster and etc. However, a patient with hand & foot fungal infections can participate.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with an American College of Rheumatology 20(ACR20) response | at baseline and week 24

SECONDARY OUTCOMES:
Proportion of patients with ACR50 response | at baseline and week 24
Proportion of patients with ACR70 response | at baseline and week 24
Mean change from baseline of Swollen joint count(SJC) and Tender joint count(TJC) respectively | at baseline and week 24
Mean change from baseline in disease activity using 28-joint modified disease activity score (DAS28) | at baseline and week 24
Proportion of patients achieving DAS28 remission (DAS28 < 2.6) | at week 24
Adverse event incidence | from baseline to week 24
Mean change from baseline to evaluation visits in vital signs | from baseline to week 24
Result of Electrocardiogram. From baseline to evaluation visits | from baseline to week 24
Mean change from baseline visit to evaluation visits in quantitative hematological exam results (including Hb, Ht, RBC, WBC & differential, platelet counts). | from baseline to week 24
Mean change from baseline visit to evaluation visits in quantitative Biochemical exam of blood results (including AST, ALT, Alk-p, γ-GTP, LDH, total protein, albumin, total bilirubin, BUN, uric acid, creatinine, glucose, ferritin, K, Na, Cl, Ca, P.). | from baseline to week 24
Mean change from baseline visit to evaluation visits in quantitative serum lipid exam results. | from baseline to week 24
Mean change from baseline visit to evaluation visits in quantitative urinalysis results. | from baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiaki Someya, Study Chair — Chugai Pharma Taiwan
Locations (12):
- Taiwan (12):
  - Buddhist Dalin Tzu Chi General Hospital, Chiayi City
  - Chang Gung Memorial Hospital -Kaohsiung, Kaohsiung City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Cathay General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan District